CLINICAL TRIAL: NCT01600274
Title: Characterisation of Relative Bioavailability and Assessment of Bioequivalence of a Newly Developed Ethinylestradiol/Dienogest IR Formulation in Comparison With a Marketed Reference Product (Valette®)
Brief Title: Bioavailability Study With Oral Single Dose Administration of Ethinylestradiol and Dienogest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharbil Waltrop GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1229ed09ct
Record Dates: First submitted 2012-05-08; First posted 2012-05-17 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Focus: Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diena (Experimental): Dienogest-Ethinyl Estradiol (test product) tablet
  Interventions: Drug: Dienogest-Ethinyl Estradiol (test product)
- Valette® (Active Comparator): Dienogest-Ethinyl Estradiol (reference product) tablet
  Interventions: Drug: Dienogest-Ethinyl Estradiol (reference product)

INTERVENTIONS:
Drug: Dienogest-Ethinyl Estradiol (test product) — One tablet of Test
  Other Names: Diena
  Arms: Diena
Drug: Dienogest-Ethinyl Estradiol (reference product) — One tablet of Reference
  Other Names: Valette®
  Arms: Valette®

SUMMARY:
* Characterisation of relative bioavailability of Diena (Test) in comparison to Valette® (Reference) after single dose administration under fasting conditions
* Assessment of bioequivalence of Test vs. Reference after single dose administration under fasting conditions, determined by use of area under the concentration time curve AUC0-tlast and maximum concentration Cmax obtained for ethinylestradiol (EE) and dienogest (DNG)
* Descriptive characterisation of safety and tolerability of the investigational products in the study population

DETAILED DESCRIPTION:
The aims of this study were to characterise relative bioavailability of Diena (Test) in comparison to Valette® (Reference) after single dose administration under fasting conditions and to assess bioequivalence of Test vs. Reference after single dose administration under fasting conditions, determined by use of area under the concentration time curve AUC0-tlast and maximal concentration Cmax obtained for ethinylestradiol (EE) and dienogest (DNG). Furthermore, a descriptive characterisation of safety and tolerability of the investigational products in the study population was performed.

ELIGIBILITY:
Inclusion Criteria:

1. sex: female
2. ethnic origin: Caucasian
3. age: 18 - 55 years, inclusive
4. body-mass index (BMI): more than 19 kg/m² and less than 27 kg/m²
5. good state of health
6. non-smoker or an ex-smoker for a least 6 months
7. written informed consent, after having been informed about benefits and potential risks of the trial, as well as details of the insurance taken out to cover the subject's participating in the study

Exclusion Criteria:

Subjects cannot be included if they match any of the following exclusion criteria:

Safety concerns

1. existing cardiac or haematological diseases and/or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
2. existing hepatic and/or renal diseases and/or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
3. existing gastrointestinal diseases and/or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
4. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
5. pathological ECG (12 standard leads) which might interfere with the safety of the active ingredient
6. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
7. subjects with severe allergies or multiple drug allergies
8. systolic blood pressure > 160 mmHg
9. diastolic blood pressure > 90 mmHg
10. heart rate < 45 and > 100 bpm
11. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the study by the investigator
12. positive anti-HIV-test, HBs-AG-test or anti-HCV-test
13. presence or history of venous or arterial thrombosis (e.g. deep venous thrombosis, pulmonary embolism, myocardial infarction and prodromal conditions (e.g. transient ischaemic attack, angina pectoris)), predisposition for venous or arterial thrombosis (e.g. APC-resistance, antithrombin-III-deficiency, protein C deficiency, protein S deficiency or other thrombogene coagulopathy, heart valve disorders or thrombogene cardiac dysrhythmias)
14. presence or history of liver tumours or known or suspected sex-hormone influenced malignancies (e.g. of the breasts or endometrium)
15. unclarified vaginal bleeding or amenorrhoe
16. subjects with fructose or galactose intolerance, deficiency of lactase, saccharase-isomaltase or malabsortion of glucose/galactose Lack of suitability for the trial
17. acute or chronic diseases which could affect absorption or metabolism
18. history of or current drug or alcohol dependence
19. regular intake of alcoholic food or beverages of ≥ 20 g per day
20. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
21. regular intake of caffeine containing food or beverages of ≥ 500 mg per day
22. blood donation or other blood loss of more than 400 ml within the last two months prior to individual enrolment of the subject
23. participation in a clinical trial during the last two months prior to individual enrolment of the subject
24. regular treatment with any systemically available medication (except usual replacement therapy with L-thyroxine)
25. subjects, who report a frequent occurrence of migraine attacks
26. use of hormonal preparations within 6 weeks (oral, transdermal, vaginal), 2 months (intramuscularly administered depot preparations used once per month) or 6 months (intramuscularly administered depot preparations used once per 3 month) before pre-study examination

    For female subjects with childbearing potential only:
27. positive pregnancy test at pre-study examination
28. pregnant or lactating women
29. female subjects who do not agree to apply adequate non-hormonal and highly effective contraceptive methods as defined in Note for Guidance on Non-Clinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceuticals (CPMP/ICH/286/95, modification), November 2000 Administrative reasons
30. subjects suspected or known not to follow instructions
31. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the study The exclusion criteria are chosen to assure that subjects with specific risks for administration of the investigated medicinal products and subjects with conditions, which may have an impact on pharmacokinetic parameters, cannot be included.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Cmax of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a.
AUC0-tlast of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a.

SECONDARY OUTCOMES:
Clast of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
AUCexpol% of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
AUC0-∞ of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
Tmax of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
t1/2 of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
tlast of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
λ of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
MRT of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a
Tlag of EE and DNG after each treatment | PK blood sampling will be performed pre-dose (within 1.5 h prior to administration) as well as 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 36, 48 and 60 h p.a

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, PhD, Principal Investigator — SocraTec R&D GmbH - Clinical Pharmacology Unit Mainzerhofplatz 14, 99084 Erfurt, Germany
Locations (1):
- SocraTec R&D, Erfurt, Thuringia, Germany